CLINICAL TRIAL: NCT01844635
Title: A Prospective Randomized Multicenter Study Comparing Different Dosages of Rabbit Antithymocyte Globulin (Thymoglobuline) in Patients With Severe Aplastic Anemia
Brief Title: Randomised Study Comparing Different Dosages of Rabbit ATG in Patients With SAA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nagoya University (Other)
Responsible Party: Principal Investigator, Hideki Muramatsu, Assistant Professor, Nagoya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APBMT AAWG-01
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Acquired Aplastic Anemia.
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2.5 mg/kg/day of Thymoglobulin for 5 days (Experimental): 2.5 mg/kg/day of Thymoglobulin for 5 days
  Interventions: Drug: Thymoglobulin
- 3.5 mg/kg/day of Thymoglobulin for 5 days (Active Comparator): 3.5 mg/kg/day of Thymoglobulin for 5 days
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin

SUMMARY:
The objective of this study is to evaluate the feasibility and effectiveness of immunosuppressive therapy (IST) using rabbit anti-thymocyte globulin (ATG) (Thymoglobuline, Genzyme) for patients with very severe aplastic anemia (VSAA) and severe aplastic anemia (SAA) as a primary therapy. The primary endpoint is the response rate (complete response (CR) + partial response (PR)) at day 180 after the start of IST. Secondary endpoints include evaluation of the presence and frequency of Epstein-Barr virus (EBV)-reactivation and EBV-associated lymphoproliferative disorder (EBV-LPD), Cytomegalovirus(CMV)-reactivation and CMV associated diseases, the response rate (CR+PR) on Day 360 after the start of IST, relapse rate and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Acquired aplastic anemia
* Age: younger than 70 years old
* Severity: SAA, VSAA.
* Interval between diagnosis and registration <6 months.
* Written informed consent from the caretakers and/or whenever possible consent from the patient.

Exclusion Criteria:

-

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Hematologic response (complete response (CR) or partial response (PR)) in patients with immunosuppressive therapy (IST) on day 180 after the start of IST. | day 180 after the start of IST

CONTACTS AND LOCATIONS:
Overall Officials: Seiji Kojima, MD., PhD., Principal Investigator — Department of Pediatrics, Nagoya University Graduate School of Medicine
Locations (1):
- Department of Pediatrics, Nagoya University Graduate School of Medicine, Nagoya, Aichi-ken, Japan